CLINICAL TRIAL: NCT00288171
Title: Randomized Double-blinded, Placebo-controlled, Cross-over Trial of Allopurinol for the Treatment of Post-renal-transplant Hypertension in Children
Brief Title: Allopurinol for Renal Transplant Associated Hypertension in Children
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: insufficient number of eligible subjects
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Baylor University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: DK64587-POST (terminated); K23DK064587 (NIH)
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Hypertension; Renal Transplant
MeSH Terms: conditions — Hypertension | interventions — Allopurinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Allopurinal (Experimental): Hypertensive renal transplant recipients with elevated uric acid will the treated with allopurinol and placebo in an randomized cross over fashion. Subjects will serve as their own controls.
  Interventions: Drug: Allopurinol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — placebo capsule twice daily for one month
  Arms: Placebo
Drug: Allopurinol — Allopurinol 200mg twice daily for one month
  Arms: Allopurinal

SUMMARY:
To test the hypothesis that lowering serum uric acid will ameliorate hypertension in children after renal transplantation.

DETAILED DESCRIPTION:
The study will be a double-blind, placebo-controlled, crossover trial. We will recruit 25 children between the ages of 6 and 18 years, from the pediatric renal transplant program at Texas Children's Hospital. The study consists of three phases, a screening phase, and a treatment phase, and a crossover phase.

Clinical study design: The study will be a double-blind, placebo-controlled, crossover trial. We will recruit 25 children between the ages of 6 and 18 years, from the pediatric renal transplant program at Texas Children's Hospital. The study consists of three phases, a screening phase, and a treatment phase, and a crossover phase.

Laboratory Measurements: The laboratory measurements will be performed in the CLIA approved, clinical laboratory at Texas Children's Hospital.

Definition of high blood pressure: We will use the guidelines for blood pressure measurement that have been adapted from the Update on the Task Force Report (1987) on High Blood Pressure in Children and Adolescents [22]. Hypertension will be defined as >95th percentile blood pressure for age, height percentile (rounded to the nearest of 5th, 10th, 25th, 50th, 75th, 90th, or 95th percentile of height above the patients actual height) and gender. Each blood pressure measurement will be the mean of 3 right arm readings, taken with an mercury sphygmomanometer at least three minutes apart with the patient sitting upright and relaxed. For the purposes of the study, to be defined as hypertensive, a patient will need to have mean systolic or diastolic blood pressure >95th percentile on three consecutive occasions, on separate days over at least a 1 week period. Patients with previously confirmed hypertension will be reconfirmed during the screening period.

Screening phase: The screening phase will last between 1 and 2 weeks. Patients will be taught to use a digital blood pressure monitor with an appropriately sized cuff and be instructed to perform daily blood pressure measurements and keep a blood pressure log. Blood tests will be done to determine eligibility based on clinical laboratory parameters. Girls who are post-menarche will have a urine pregnancy test. Each child will undergo 24hr ambulatory blood pressure monitoring during the screening phase. Children will collect urine for 24-hours for the purpose of screening urinary nitrates and bradykinin.

Phase 1: The active phase will last six weeks and include a clinic visit on the first day of the phase, laboratory testing between day 4 and 7, and weekly telephone contact throughout the phase. Subjects will receive allopurinol or placebo. Laboratory tests will be performed 4 to 7 days after starting the medication to screen for hepatic or bone marrow toxicity (AST, ALT, CBC), renal function (Cr), cyclosporin or tacrolimus level and serum uric acid. Evidence for toxicity, increased creatinine or unstable cyclosporin levels will lead to immediate discontinuation of allopurinol withdrawal from the study. The families will also be instructed to continue the daily blood pressure log started in the screening phase. At the end of the phase, prior to discontinuation of the allopurinol, children will again undergo 24hr ambulatory blood pressure monitoring. Children will repeat the 24-hour urine collection for the purpose of screening urinary nitrates and bradykinin.

Washout Phase: There will be a two-week washout interval between the allopurinol and placebo phases.

Crossover Phase: The crossover phase will identical in procedures to the active phase except that the children will be receiving allopurinol or placebo, whichever was not received in Phase 1.

ELIGIBILITY:
Inclusion Criteria:

Males or females 6 to 18 years in age. Post-menarche females must have a negative urine pregnancy test.

Renal transplant recipient taking cyclosporin.

Weight greater than 20kg

Parental or guardian consent and child subject assent (if appropriate)

SBP or DBP greater than 95th percentile for age, gender and height

Exclusion Criteria:

Severe or poorly controlled hypertension as defined by SBP or DBP more than 20mmHg >95th percentile for age, gender and height on active therapy, on 2 or more antihypertensive medications or a history of hypertensive encephalopathy

Taking azathioprine or another nucleoside analogue medication

Currently receiving ACE-I or ARB medications

Laboratory abnormalities that indicate clinically significant hematologic, hepatobiliary or renal disease: Schwartz Formula GFR less than 60ml/min/1.73m2 ALT/SGPT greater than 2 times the upper limit of normal* Hemoglobin less than 9 gm/dl WBC less than 3.000/mm3 Platelet count less than 100,000/mm3 *age-adjusted normal range, TCH laboratory

A history of cardiomyopathy, clinically significant structural heart disease or atrioventricular conduction disturbance, sick sinus syndrome, clinically significant cardiac arrhythmia or symptoms of congestive heart failure

Pregnant or lactating females

Any other investigational drug use within 30 days of enrollment

Parents/guardians or subjects who, in the opinion of the investigator, may be non-compliant with the study procedures.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2006-02; Primary Completion 2008-01 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Systolic Blood Pressure | 2 months

SECONDARY OUTCOMES:
Serum Creatinine | 2 months
urinary bradykinin | 2 months
urinary nitrates | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel I Feig, MD, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States